CLINICAL TRIAL: NCT02114294
Title: Does Isolated Hip Strengthening for Patellofemoral Pain Syndrome Give Better Long Term Results Than Traditional Quadriceps Based Training? A Randomised Controlled Trial.
Brief Title: Hip Strengthening Versus Quadriceps Based Training for Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/1860REK
Record Dates: First submitted 2014-02-14; First posted 2014-04-15 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrome; Anterior knee pain; Randomised controlled trial; Exercise intervention; Hip strengthening; Quadriceps based training; Anterior knee pain score
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isolated hip strengthening (Experimental): Isolated hip strengthening (abduction, external rotation, extension)
  Interventions: Other: Isolated hip strengthening
- Quadriceps based training (Active Comparator): Quadriceps based training (mini-squat, straight leg raising, terminal extensions)
  Interventions: Other: Quadriceps based training
- Active control (Other): Patients receive standardised information concerning patellofemoral pain syndrome, but receive no prescribed exercise regime. They are encouraged to remain active.
  Interventions: Other: Active control

INTERVENTIONS:
Other: Isolated hip strengthening — Exercise program that is carried out by subjects under supervision once a week and then performed at home 2 additional times without supervision for a total of 6 weeks. Hip strengthening group will train hip abduction, hip external rotation and hip extension.
  Arms: Isolated hip strengthening
Other: Quadriceps based training — Exercise program that is carried out by subjects under supervision once a week and then performed at home 2 additional times without supervision for a total of 6 weeks. Quadriceps group will train mini-squat, straight leg raising, terminal extensions.
  Arms: Quadriceps based training
Other: Active control — Patients receive standardised information concerning patellofemoral pain syndrome, but receive no prescribed exercise regime. They are encouraged to remain active.
  Arms: Active control

SUMMARY:
This is a Randomized Controlled Trial (RCT) regarding conservative treatment of Patellofemoral Pain Syndrome (PFPS). Patellofemoral Pain Syndrome (PFPS) is a very common cause of knee pain in young active adults with a high rate of recurrent and/or chronic occurrence. PFPS is notoriously difficult to treat and has been referred to as "one of the most vexatious clinical challenges in rehabilitative medicine". Its etiology is unclear but is commonly thought to be related to pathomechanics in the patellofemoral joint (PFJ). There are many factors that can influence PFJ mechanics. Among these, quadriceps strength and timing has been shown to be important. As such, treatment of PFPS has traditionally been based on correction of pathomechanics through influencing quadriceps strength and timing. However, a growing body of evidence is revealing the importance of strength and control of hip abduction and external rotation in PFPS. Hip strength in ab/adduction and rotation is thought to influence femoral positioning in the patellofemoral joint, thereby affecting PFJ mechanics. Several cohort and smaller RCT studies within the last 7 years have shown that additional exercises for hip strength and control give an improved effect in pain and function compared with quadriceps based training alone. A smaller RCT from 2012 compared isolated hip strengthening exercises to a control group and found surprisingly good results on pain in function in the hip strengthening group. The investigators plan a RCT in which isolated hip strengthening will be compared to traditional quadriceps training and a control group which will receive no structured training. Primary outcomes will be pain and function. This high-quality study will include 40-50 patients in each group, making it one of the largest of its kind on conservative treatment for PFPS. In contrast to the vast majority of studies of this type, this study will also include men, which will potentially help to fill a significant gap in the literature on this subject. The investigators study will therefore be an important contribution to elucidating the etiology of PFPS and improving treatment options for both men and women in the future. As well, the role of psychometric parameters will be examined and a standardized clinical test for hip abduction endurance will be developed. Follow-up at 3 months and 12 months is completed and published. A 5-year follow-up of the same patients is underway.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-40 years
* Insidious onset of symptoms not related to trauma
* Symptoms more than 3 months
* A minimum of VAS 3 on VAS-W
* Peri- or retropatellar pain during or after at least two of the following: Stair ascent or descent, hopping, running, prolonged sitting, squatting, kneeling.
* Pain on one of the following: Compression of the patella, palpation of the patellar facets

Exclusion Criteria:

* Clinical findings indicative of meniscal or other intraarticular injury
* Clinical findings indicative of injury to or increased laxity of cruciate or collateral ligaments
* Findings on MRI indicative of other intraarticular pathology.
* Clinical and/or x-ray findings (plain anterior-posterior, lateral and skyline view) indicative of osteoarthritis, Osgood-Schlatter or Sinding-Larsen-Johanssen syndrome
* Clinical findings indicative of knee joint effusion
* Significant pain from hip or lumbar spine on clinical evaluation, with potential for causing referred pain to the knee or hindering the patient's ability to perform the prescribed exercises.
* Recurrent patellar subluxation or dislocation.
* Previous surgery to the knee joint
* NSAID or cortisone use over an extended period of time
* Having suffered trauma to the knee joint judged during clinical evaluation to have a significant effect on the presenting clinical condition.
* Physiotherapy or other similar treatment for patellofemoral pain syndrome within the previous 3 months

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Anterior knee pain score | 3 months
  Anterior Knee Pain Score (AKPS) is a measurement of subjective symptoms and functional limitations in patellofemoral pain, and has been validated for use in this patient population. The AKPS consists of a 13-point questionnaire with categories related to different levels of function in the knee. The categories within each question are weighted, and the responses are summed for an overall index where 100 represents perfect function. The mean clinically important difference (MCID) has been determined to be 10 points. This questionnaire will be translated to Norwegian and validated according to standard scientific procedures with approval from Kuala et al.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 3 months
  Visual Analog Scale (VAS) for pain (0-10cm)
Global Score Global Score | 3 months
  An 18-point likert scale for measuring patients' global assessment of change compared with baseline will be carried out at 3 and 12 months. The scale ranges from -9 (maximum deterioration) to +9 (maximum improvement).
Step-down test | 3 months
  The step down as performed according to standardised instruction will be used to quantify changes in patients' function. The measure is number of repetitions in 30 seconds.
Hip abduction, external rotation and knee extension strength | 3 months
  Isometric strength will be measured for hip abduction, hip external rotation and knee extension.
Hip abduction endurance | 3 months
  Testing is carried out in side-lying position with a 5kg weight around the ankle of the upper leg, which is abducted to 30 degrees above the horizontal plane. Time successfully held in target area is measured in seconds.
EQ 5D 5L | 3 months
  EQ-5D-5L is calculated on the basis of five questions about daily activities, pain and psychological status with five possible answers for each question. In addition the subject scores his/her overall health on a 1-100 scale. The results are translated to a single summary index value through the use of a table
Tampa scale for kinesiophobia | 3 months
  The Tampa scale for kinesiophobia (TSK) is a 13 -item questionnaire aimed at the assessment of fear of movement/re-injury. Each item is scored on a 4-point Likert scale with alternatives ranging from "strongly disagree" (0) to "strongly agree". This gives a possible total score range from 0 to 52.
HSCL-10 | 3 months
  The Hopkins Symptom Checklist (HSCL) is a symptom inventory which measures symptoms of anxiety and depression.
Knee self-efficacy score (K-SES) | 3 months
  K-SES is a self-administered instrument consisting of in total four sections in which patients score how certain they are about specific activities currently and in the future.
Pain drawing with number of painful regions | 3 months
  An adaptation of the Standardised Nordic Questionnaire will be used to register the number of painful areas.

CONTACTS AND LOCATIONS:
Overall Officials: Sigurd Liavaag, MD, PhD, Study Director — Sørlandet sykehus HF; Alexandra C Hott, MD, Principal Investigator — Sørlandet sykehus HF
Locations (1):
- Sorlandet hospital, Kristiansand, Vest Agder, Norway

REFERENCES:
- [Background] Witvrouw E, Werner S, Mikkelsen C, Van Tiggelen D, Vanden Berghe L, Cerulli G. Clinical classification of patellofemoral pain syndrome: guidelines for non-operative treatment. Knee Surg Sports Traumatol Arthrosc. 2005 Mar;13(2):122-30. doi: 10.1007/s00167-004-0577-6. Epub 2005 Feb 10. PMID 15703965
- [Background] Witvrouw E, Danneels L, Van Tiggelen D, Willems TM, Cambier D. Open versus closed kinetic chain exercises in patellofemoral pain: a 5-year prospective randomized study. Am J Sports Med. 2004 Jul-Aug;32(5):1122-30. doi: 10.1177/0363546503262187. Epub 2004 May 18. PMID 15262632
- [Background] Souza RB, Draper CE, Fredericson M, Powers CM. Femur rotation and patellofemoral joint kinematics: a weight-bearing magnetic resonance imaging analysis. J Orthop Sports Phys Ther. 2010 May;40(5):277-85. doi: 10.2519/jospt.2010.3215. PMID 20436239
- [Background] Khayambashi K, Mohammadkhani Z, Ghaznavi K, Lyle MA, Powers CM. The effects of isolated hip abductor and external rotator muscle strengthening on pain, health status, and hip strength in females with patellofemoral pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):22-9. doi: 10.2519/jospt.2012.3704. Epub 2011 Oct 25. PMID 22027216
- [Background] Dolak KL, Silkman C, Medina McKeon J, Hosey RG, Lattermann C, Uhl TL. Hip strengthening prior to functional exercises reduces pain sooner than quadriceps strengthening in females with patellofemoral pain syndrome: a randomized clinical trial. J Orthop Sports Phys Ther. 2011 Aug;41(8):560-70. doi: 10.2519/jospt.2011.3499. Epub 2011 Jun 7. PMID 21654093
- [Background] Fukuda TY, Melo WP, Zaffalon BM, Rossetto FM, Magalhaes E, Bryk FF, Martin RL. Hip posterolateral musculature strengthening in sedentary women with patellofemoral pain syndrome: a randomized controlled clinical trial with 1-year follow-up. J Orthop Sports Phys Ther. 2012 Oct;42(10):823-30. doi: 10.2519/jospt.2012.4184. Epub 2012 Aug 2. PMID 22951491
- [Background] Nakagawa TH, Muniz TB, Baldon Rde M, Dias Maciel C, de Menezes Reiff RB, Serrao FV. The effect of additional strengthening of hip abductor and lateral rotator muscles in patellofemoral pain syndrome: a randomized controlled pilot study. Clin Rehabil. 2008 Dec;22(12):1051-60. doi: 10.1177/0269215508095357. PMID 19052244
- [Background] Prins MR, van der Wurff P. Females with patellofemoral pain syndrome have weak hip muscles: a systematic review. Aust J Physiother. 2009;55(1):9-15. doi: 10.1016/s0004-9514(09)70055-8. PMID 19226237
- [Background] Kujala UM, Jaakkola LH, Koskinen SK, Taimela S, Hurme M, Nelimarkka O. Scoring of patellofemoral disorders. Arthroscopy. 1993;9(2):159-63. doi: 10.1016/s0749-8063(05)80366-4. PMID 8461073
- [Derived] Hott A, Pripp AH, Juel NG, Liavaag S, Brox JI. Self-efficacy and Emotional Distress in a Cohort With Patellofemoral Pain. Orthop J Sports Med. 2022 Mar 8;10(3):23259671221079672. doi: 10.1177/23259671221079672. eCollection 2022 Mar. PMID 35284585
- [Derived] Hott A, Brox JI, Pripp AH, Juel NG, Liavaag S. Predictors of Pain, Function, and Change in Patellofemoral Pain. Am J Sports Med. 2020 Feb;48(2):351-358. doi: 10.1177/0363546519889623. Epub 2019 Dec 10. PMID 31821014
- [Derived] Hott A, Liavaag S, Juel NG, Brox JI, Ekeberg OM. The reliability, validity, interpretability, and responsiveness of the Norwegian version of the Anterior Knee Pain Scale in patellofemoral pain. Disabil Rehabil. 2021 Jun;43(11):1605-1614. doi: 10.1080/09638288.2019.1671499. Epub 2019 Oct 4. PMID 31583918
- [Derived] Hott A, Brox JI, Pripp AH, Juel NG, Paulsen G, Liavaag S. Effectiveness of Isolated Hip Exercise, Knee Exercise, or Free Physical Activity for Patellofemoral Pain: A Randomized Controlled Trial. Am J Sports Med. 2019 May;47(6):1312-1322. doi: 10.1177/0363546519830644. Epub 2019 Apr 8. PMID 30958707
- [Derived] Hott A, Liavaag S, Juel NG, Brox JI. Study protocol: a randomised controlled trial comparing the long term effects of isolated hip strengthening, quadriceps-based training and free physical activity for patellofemoral pain syndrome (anterior knee pain). BMC Musculoskelet Disord. 2015 Feb 25;16:40. doi: 10.1186/s12891-015-0493-6. PMID 25879452